CLINICAL TRIAL: NCT01211470
Title: Randomized, Dose Ranging, Active Controlled Efficacy and Safety Evaluation of PMX-30063 As Initial Treatment for Acute Bacterial Skin and Skin Structure Infections (ABSSSI) Caused by Staphylococcus Aureus
Brief Title: Initial Treatment for Acute Bacterial Skin Infections (ABSSSI) Caused by Staphylococcus Aureus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PolyMedix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PROTOCOL PMX63-203
Record Dates: First submitted 2010-09-27; First posted 2010-09-29 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: Acute Bacterial Skin and Skin-structure Infection(ABSSSI) Due to Staphylococcus Aureus (MSSA); (Susceptible or Methicillin Resistant)
Keywords: MRSA; ABSSSI; Staphylococcus aureus
MeSH Terms: conditions — Disease Susceptibility; Staphylococcal Infections | interventions — Daptomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PMX-30063 (Experimental): 3 arms of PMX-300063
  Interventions: Drug: PMX-30063-investigational drug
- Daptomycin. (Active Comparator): Daptomycin will be administered according to the approved product monograph information for ABSSSI.
  Interventions: Drug: Daptomycin

INTERVENTIONS:
Drug: Daptomycin — Active Comparator: Daptomycin.
  Arms: Daptomycin.
Drug: PMX-30063-investigational drug — Experimental: PMX-30063
  Arms: PMX-30063

SUMMARY:
The study investigates the safety and efficacy of PMX-30063 in patients treated for acute bacterial skin and skin-structure infection (ABSSSI).

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of ABSSSI in which S. aureus is clinically suspected to be the likely pathogen
2. Clinical manifestation of subjects' ABSSSI must include the presence of purulent material suitable for microbiologic culture, Gram stain examination and PCR assay.
3. The ABSSSI must be 75 cm2 or greater in size in order for the subject to be eligible for this study. This includes the primary and surrounding erythema, swelling or induration.
4. Super-infected eczema or other chronic medical conditions (e.g., atopic dermatitis, hidradentitis suppurativa) characterized by prominent signs of inflammation for an extended period even after successful bacterial eradication. (Subjects with an ABSSSI that involves an anatomic location in which there is no evidence of a chronic skin condition are eligible for enrollment.)

Exclusion Criteria:

1. Female patients who are pregnant, lactating (breast milk feeding), or planning a pregnancy during the course of the study.
2. History of peripheral neuropathy of any form or etiology
3. Anticipated need for prolonged antibiotic therapy (i.e., >8 days)
4. ABSSSI known or suspected to be caused exclusively by Gram negative pathogens or anaerobes (both Gram positive or Gram negative)
5. Diabetic foot infection: defined as a subacute or chronic infection (> 4 weeks) below the ankle in a patient with diabetic neuropathy
6. Infected burns
7. Known infection with human immunodeficiency virus (HIV) and a CD4 count < 200/mm3
8. Active hepatitis B or hepatitis C receiving treatment with interferon or other immunosuppressive therapy

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The Primary objective of this study is to assess the efficacy of PMX-30063 in patients treated for acute bacterial skin and skin-structure infection (ABSSSI). | Eradication at end of treatment (day 7/8)
  The Primary objective of this study is to assess the efficacy of PMX-30063 in patients treated for acute bacterial skin and skin-structure infection (ABSSSI). The primary measure of efficacy will be bacteriologic eradication at end of treatment of S. aureus (either Methicillin-susceptible (MSSA) or Methicillin-resistant (MRSA)) in subjects with ABSSSI and having S. aureus isolated from an appropriate infection site prior to randomization.
  The secondary objectives are clinical responses, safety and pharokinetics of PMX-300063.

CONTACTS AND LOCATIONS:
Locations (8):
- Canada (6):
  - Hamilton, Ontario
  - Chicoutimi, Quebec
  - Greenfield Park, Quebec
  - Québec, Quebec
  - Sherbrooke, Quebec
  - Trois-Rivières, Quebec
- 11 Sites, Multiple, Russia
- 5 Sites, Multiple, Ukraine